CLINICAL TRIAL: NCT05829005
Title: Trial of Neurostimulation Treatment and Investigation for Causes of Functional Motor Symptoms: a Pilot Study
Acronym: TONICS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: South London and Maudsley NHS Foundation Trust (Other); King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 250915
Record Dates: First submitted 2023-01-16; First posted 2023-04-25 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Functional Neurological Symptom Disorder
Keywords: Functional neurological disorder
MeSH Terms: conditions — Conversion Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Multi-centre, two-arm (active TMS, inactive TMS), double-blind (outcome assessor, patient), parallel-group RCT. Patients and researchers rating outcomes will be blind to the treatment arm, but it is not possible to blind the (different) researcher who is administering the treatments.
  There will be two treatment sessions, between 4-20 days apart, and two follow-up assessments one and three months after the first treatment session.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active arm (Active Comparator): The location and number of pulses will be set. The intensity of stimulation will be felt by the subject. 120 stimuli - including at least 20 supra (motor) threshold stimuli causing movement of the affected limb.
  Interventions: Device: Transcranial magnetic stimulation (TMS)
- Inactive/control arm (Sham Comparator): The location and number of pulses have been set at the same as the active treatment. The intensity of stimulation will necessarily be less but will still result in a stimulus that is felt by the subject to maximise chances of successful blinding. 120 stimuli - no stimuli of sufficient intensity to produce movement.
  Interventions: Device: Transcranial magnetic stimulation (TMS)

INTERVENTIONS:
Device: Transcranial magnetic stimulation (TMS) — TMS is a form of 'non-invasive brain stimulation', i.e. it is a way of stimulating the brain from outside the head. It works by holding a magnetic coil approximately the size of a small side plate against the head (it rests on the scalp) which then delivers magnetic pulses that stimulate the underlying brain. It was developed over 30 years ago and has been increasingly used to treat a number of neurological and psychiatric disorders. It is considered a relatively safe and generally well-tolerated treatment.

SUMMARY:
A pilot randomised controlled trial (RCT) of single-pulse transcranial magnetic stimulation (TMS) over the motor cortex to investigate efficacy in improving motor FND symptoms and to make a preliminary investigation of predictors of response to TMS and potential mechanisms of action.

DETAILED DESCRIPTION:
This study is a pilot trial that will aim to determine if Transcranial Magnetic Stimulation (TMS) is an effective, tolerated and safe treatment for functional neurological disorder (FND) and to make a preliminary investigation of predictors of response to TMS and potential mechanisms of action.

This trial will be a 'randomised, two-arm, double-blind, parallel-arm study design. Randomised means that patients will be allocated to 'active' or 'inactive' treatment groups at random - this is done to minimise the chances of the characteristics of groups being different and influencing response to the different treatments. Double-blind means that the patients will not know which group they have been allocated to, and the assessors of response to treatment will be blinded, which will help reduce researcher 'bias' in assessing response. Parallel means that the treatment groups will occur alongside each other and patients will only have one of the treatments during the trial - unlike a 'crossover' design where patients will get both. However, after the trial, if a patient has received the 'inactive' treatment they will be offered the 'active' treatment if, after review by the clinician, such treatment is considered appropriate by the clinician.

The 'active' intervention is supra-threshold TMS that is so-called as it above the threshold needed to stimulate the primary motor cortex, the area of the brain known as 'M1' that when stimulated leads to contraction of limb muscles and can therefore make a weak limb move that the patient would otherwise not be able to move. This study postulates that it is the stimulation of a paralysed limb resulting in movement that is the active component of treatment, as it allows patients to relearn and re-experience normal movement, as well as providing proof of the possibility of the return of function.

An 'inactive' control arm is being used in this study as this is the standard way to show if, and how much, any response to the 'active' intervention might be due to chance. The investigators will be using sub-threshold TMS, so real TMS that will stimulate the motor cortex. This is different to other options for the control arm, such 'sham' TMS where no actual TMS pulse is delivered. Such sham devices deliver a similar sensation to the scalp and are designed to look the same as 'real' TMS devices so it is hard, and ideally impossible, for the patient to know whether they were getting real or sham treatment. This will also be delivered to the same location (primary motor cortex, ie. 'M1'). The location and number of pulses have been set at the same as the active treatment. The intensity of stimulation will necessarily be less, but will still result in a stimulus that is felt by the subject to maximise chances of successful blinding.

Importantly, and necessarily, details of what the two arms will involve are kept vague in the information sheet to maximise the chances of successful blinding of participants. There is genuine equipoise between these two proposed arms because, as yet, there is no evidence that the reported effects of TMS in the published case series are anything other than placebo. The one published feasibility RCT found no significant increase in subjective ratings of strength compared to placebo.

The use of blinded assessments of some clinician-rated measures and use of patient-rated outcomes (including the primary outcome measure) will reduce "researcher effects" and "researcher bias", as will use of the local (KCL) clinical trials unit (CTU) database system. During the trial, any changes in other treatments will be carefully documented at the start of treatment and at all subsequent assessments. No attempt will be made to standardise these or balance them between the arms other than randomisation but the effects of these, and other pertinent changes (e.g. other clinical parameters such as anxiety and depression scores) to see if they mediate outcomes.

Timetable

The research project will take approximately 12 months to complete after ethical approval. The investigators aim to randomise 60 patients to one of the treatment arms. The investigators anticipate being able to recruit at a rate of approximately 3 per week, therefore taking 20 weeks (5 months) to complete recruitment. This can be rounded up to 7 months to allow for slow initial recruitment whilst recruitment pathways are set up and for possible initial delays in starting first patients due to arranging mutually convenient times for consenting, assessing and first treatment session. Each patient will then take 5 months to complete the study, so the last patients will finish follow up 12 months after the first patient is recruited. There are no planned interim analyses/reports.

Study details

Recruitment

This will be from inpatient and outpatient settings in London.

The neuropsychiatry services of King's Health Partners (KHP). KHP is an Academic Health Sciences Centre comprising the National Health Service (NHS) Foundation Trusts associated with King's College London (KCL) directly serving 2 million patients in South East London. KHP has two regional neurosciences centres at King's College Hospital (KCH) and St.Thomas'/Guys Hospitals NHS foundation trusts. They will also be recruited from South West London & St George's Mental Health NHS Trust (SWLSTG) and University College London Hospitals NHS Foundation Trust (UCLH). The South London and Maudsley NHS Foundation Trust (SLaM) is the UK's largest Mental Health Trust. All 3 trusts receive many FND referrals from the local population but also from the South East of England and beyond. Assessments will be in private rooms at the relevant hospitals or the Institute of Psychiatry, Psychology and Neuroscience (IoPPN - a faculty of KCL at the Denmark Hill campus next to KCH and Maudsley Hospitals). TMS treatments will be in specialist treatment rooms either at KCH (department of neurophysiology) or IoPPN (department of psychosis studies).

Suitable patients will be identified by the clinical team involved in their care who will inform them about the study and either give them directly (in the clinic or on the ward) or send them by post, the information sheet about the study and invite them to get in touch with a member of the research team as detailed in the information sheet. If the patient is seen face-to-face by the clinician they will ask if the patient is willing for their details to be passed on to the research team so they can contact them directly by their preferred method of contact (post, phone or email). If the patient is sent an information sheet they will be told they will receive a phone call following up the letter within 2 weeks of receiving it to enquire as to whether they are interested in taking part, with reassurance that there will be no further contact from the research team if they do not wish to find out more about the study which they can convey to the research team when called on the phone (or do beforehand by contacting the research team via mail, email or phone)

60 patients are widely considered a standard sample for such a pilot study.

Patient visits, assessments and treatments:

The full project protocol (attached to this application), and later sections of this form, give full details of the timing of visits/participants' potential flow through the study, assessment forms/measures and the technical specifications of the treatments.

In summary, 60 patients will undergo a maximum of 5 visits to the Denmark Hill campus (with an approximate length of time of visit):

Visit A - for Screening +/- consent (15 minutes) Visit B - for Consent (if not already done) / Baseline assessments (2 hours) Visit C - for 1st Treatment session + pre & post-treatment assessments (2 hours) Visit D - for 2nd Treatment session + pre & post-treatment assessments (2 hours) Visit E - for 1st (interim) follow up for outcome assessment (1-2 hours) Visit F - for 2nd (final) follow up assessment (1-2 hours)

Visit A could be conducted by phone (and consent delayed to visit B) or combined with visit B to suit patient preference and the circumstances of recruitment. Visits E and F could be carried out as home visits or by telephone as required.

The start of treatment (visit C) will be a maximum of 2 weeks after Baseline assessments (visit B) and randomisation will take place immediately before the first treatment session. The 2nd treatment (visit D) is between 4-20 days after the 1st treatment (visit C). The follow-up assessments (visits D and E) are 1 and 3 months after the 1st treatment session (visit C).

Some assessments, such as those covering fixed characteristics (e.g. demographics) or historical details (e.g. medical, psychiatric and treatment history) will be performed only once at baseline. Other assessments such as symptoms and other changeable characteristics will be performed serially. See protocol for full details.

Both treatment arms involved delivering 120 singles pules of TMS with a circular coil to the motor cortex (M1), the first 100 of which will be used to determine motor threshold (MT) but not generate twitch of any muscle that can be seen or felt by the patient. For the active arm, the final 20 pulses will be 'supra-motor threshold' (120% of MT) in that they will cause a palpable contraction of the muscles and a visible movement of the weak limb that is confirmed by the patient. For the inactive arm, these final 20 pulses will be a 'sub-motor threshold' (80% of MT) that won't cause a palpable or visible contraction of the weak limb. No specific suggestion of recovery will be used in either arm beyond that inherent in a trial of a novel therapy - i.e. no 'enhancement' of the placebo effect will be utilised.

At the end of the final follow up patients will be unblinded and a full debrief will be given by the PI. If they were in the inactive treatment arm the possibility of receiving sessions of active treatment will be discussed with them - and if the patient and the clinician both agree this indicated it will then be offered to the patient.

ELIGIBILITY:
Inclusion Criteria

1. The Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) diagnosis of motor FND (i.e. presenting with weakness of at least one limb) made by consultant neurologist and/or neuropsychiatrist.
2. Age ≥18yrs.
3. Ability to give written informed consent.

Exclusion Criteria

1. Epilepsy (or considered high risk of epilepsy from medical history).
2. Other contraindication to TMS (e.g. cochlear implants, metallic intracranial clips/surgery in last 12 months).
3. Comorbid organic neurological condition.
4. Pain as primary symptom.
5. Previous treatment with TMS (for any condition).
6. Non-fluent English speakers (if unable to accurately complete self-report questionnaires).
7. Major mental health disorder: current diagnosis of schizophrenia or bipolar disorder; current drug/alcohol dependence.
8. History of factitious disorder.
9. Currently involved in another trial.
10. Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Adapted Patient Clinical Global Impression of Improvement (CGI-I) scale | immediately before treatment 1
  Adapted Patient Clinical Global Impression of Improvement (CGI-I) scale rated by the patient is a 7-point scale of improvement from 'very much improved' to 'very much worse'. 'Very much improved' means a better outcome.
Adapted Patient Clinical Global Impression of Improvement (CGI-I) scale | immediately after treatment 1
  Adapted Patient Clinical Global Impression of Improvement (CGI-I) scale rated by the patient is a 7-point scale of improvement from 'very much improved' to 'very much worse'. 'Very much improved' means a better outcome.
Adapted Patient Clinical Global Impression of Improvement (CGI-I) scale | immediately before treatment 2
  Adapted Patient Clinical Global Impression of Improvement (CGI-I) scale rated by the patient is a 7-point scale of improvement from 'very much improved' to 'very much worse'. 'Very much improved' means a better outcome.
Adapted Patient Clinical Global Impression of Improvement (CGI-I) scale | immediately after treatment 2
  Adapted Patient Clinical Global Impression of Improvement (CGI-I) scale rated by the patient is a 7-point scale of improvement from 'very much improved' to 'very much worse'. 'Very much improved' means a better outcome.
Adapted Patient Clinical Global Impression of Improvement (CGI-I) scale | one-month follow-up
  Adapted Patient Clinical Global Impression of Improvement (CGI-I) scale rated by the patient is a 7-point scale of improvement from 'very much improved' to 'very much worse'. 'Very much improved' means a better outcome.
Adapted Patient Clinical Global Impression of Improvement (CGI-I) scale | three-month follow-up
  Adapted Patient Clinical Global Impression of Improvement (CGI-I) scale rated by the patient is a 7-point scale of improvement from 'very much improved' to 'very much worse'. 'Very much improved' means a better outcome.

SECONDARY OUTCOMES:
Adapted Outcome Assessor Clinical Global Impression of Improvement (CGI-I) scale | immediately before treatment 1
  Adapted Patient Clinical Global Impression of Improvement (CGI-I) scale rated by the outcome assessor is a 7-point scale of improvement from 'very much improved' to 'very much worse'. 'Very much improved' means a better outcome.
Adapted Outcome Assessor Clinical Global Impression of Improvement (CGI-I) scale | immediately after treatment 1
  Adapted Patient Clinical Global Impression of Improvement (CGI-I) scale rated by the outcome assessor is a 7-point scale of improvement from 'very much improved' to 'very much worse'. 'Very much improved' means a better outcome.
Adapted Outcome Assessor Clinical Global Impression of Improvement (CGI-I) scale | immediately before treatment 2
  Adapted Patient Clinical Global Impression of Improvement (CGI-I) scale rated by the outcome assessor is a 7-point scale of improvement from 'very much improved' to 'very much worse'. 'Very much improved' means a better outcome.
Adapted Outcome Assessor Clinical Global Impression of Improvement (CGI-I) scale | immediately after treatment 2
  Adapted Patient Clinical Global Impression of Improvement (CGI-I) scale rated by the outcome assessor is a 7-point scale of improvement from 'very much improved' to 'very much worse'. 'Very much improved' means a better outcome.
Adapted Outcome Assessor Clinical Global Impression of Improvement (CGI-I) scale | one-month follow-up
  Adapted Patient Clinical Global Impression of Improvement (CGI-I) scale rated by the outcome assessor is a 7-point scale of improvement from 'very much improved' to 'very much worse'. 'Very much improved' means a better outcome.
Adapted Outcome Assessor Clinical Global Impression of Improvement (CGI-I) scale | three-month follow-up
  Adapted Patient Clinical Global Impression of Improvement (CGI-I) scale rated by the outcome assessor is a 7-point scale of improvement from 'very much improved' to 'very much worse'. 'Very much improved' means a better outcome.
Adapted Carer Clinical Global Impression of Improvement (CGI-I) scale | immediately before treatment 1
  Adapted Patient Clinical Global Impression of Improvement (CGI-I) scale rated by the carer is a 7-point scale of improvement from 'very much improved' to 'very much worse'. 'Very much improved' means a better outcome.
Adapted Carer Clinical Global Impression of Improvement (CGI-I) scale | immediately after treatment 1
  Adapted Patient Clinical Global Impression of Improvement (CGI-I) scale rated by the carer is a 7-point scale of improvement from 'very much improved' to 'very much worse'. 'Very much improved' means a better outcome.
Adapted Carer Clinical Global Impression of Improvement (CGI-I) scale | immediately before treatment 2
  Adapted Patient Clinical Global Impression of Improvement (CGI-I) scale rated by the carer is a 7-point scale of improvement from 'very much improved' to 'very much worse'. 'Very much improved' means a better outcome.
Adapted Carer Clinical Global Impression of Improvement (CGI-I) scale | immediately after treatment 2
  Adapted Patient Clinical Global Impression of Improvement (CGI-I) scale rated by the carer is a 7-point scale of improvement from 'very much improved' to 'very much worse'. 'Very much improved' means a better outcome.
Adapted Carer Clinical Global Impression of Improvement (CGI-I) scale | one-month follow-up
  Adapted Patient Clinical Global Impression of Improvement (CGI-I) scale rated by the carer is a 7-point scale of improvement from 'very much improved' to 'very much worse'. 'Very much improved' means a better outcome.
Adapted Carer Clinical Global Impression of Improvement (CGI-I) scale | three-month follow-up
  Adapted Patient Clinical Global Impression of Improvement (CGI-I) scale rated by the carer is a 7-point scale of improvement from 'very much improved' to 'very much worse'. 'Very much improved' means a better outcome.
Strength patient ratings | immediately before treatment 1
  Strength ratings assessed by the patient is a 5-point scale of strength from 'No weakness at all' to 'Very severe weakness'. 'No weakness at all' means a better outcome.
Strength patient ratings | immediately after treatment 1
  Strength ratings assessed by the patient is a 5-point scale of strength from 'No weakness at all' to 'Very severe weakness'. 'No weakness at all' means a better outcome.
Strength patient ratings | immediately before treatment 2
  Strength ratings assessed by the patient is a 5-point scale of strength from 'No weakness at all' to 'Very severe weakness'. 'No weakness at all' means a better outcome.
Strength patient ratings | immediately after treatment 2
  Strength ratings assessed by the patient is a 5-point scale of strength from 'No weakness at all' to 'Very severe weakness'. 'No weakness at all' means a better outcome.
Strength patient ratings | one-month follow-up
  Strength ratings assessed by the patient is a 5-point scale of strength from 'No weakness at all' to 'Very severe weakness'. 'No weakness at all' means a better outcome.
Strength patient ratings | three-month follow-up
  Strength ratings assessed by the patient is a 5-point scale of strength from 'No weakness at all' to 'Very severe weakness'. 'No weakness at all' means a better outcome.
Dynamometer | immediately before treatment 1
  Strength ratings measured by dynamometer
Dynamometer | immediately after treatment 1
  Strength ratings measured by dynamometer
Dynamometer | immediately before treatment 2
  Strength ratings measured by dynamometer
Dynamometer | immediately after treatment 2
  Strength ratings measured by dynamometer
Dynamometer | one-month follow-up
  Strength ratings measured by dynamometer
Dynamometer | three-month follow-up
  Strength ratings measured by dynamometer
Change from baseline computerised attention tasks | one-month follow-up
  attention task will be tested using a computer
Change from baseline computerised sense of agency tasks | one-month follow-up
  sense of agency tasks will be tested using computer
EuroQol 5-Dimension 5-Level (EQ-5D-5L) | immediately before treatment 1
  EuroQol 5-Dimension 5-Level (EQ-5D-5L), is the 5-digit code measuring functional ability. Each dimension in the EQ-5D-5L has five response levels: no problems (Level 1); slight; moderate; severe; and extreme problems (Level 5). There are 3,125 possible health states defined by combining one level from each dimension, ranging from 11111 (full health) to 55555 (worst health). A lower score means a better outcome.
EuroQol 5-Dimension 5-Level (EQ-5D-5L) | one-month follow-up
  EuroQol 5-Dimension 5-Level (EQ-5D-5L), is the 5-digit code measuring functional ability. Each dimension in the EQ-5D-5L has five response levels: no problems (Level 1); slight; moderate; severe; and extreme problems (Level 5). There are 3,125 possible health states defined by combining one level from each dimension, ranging from 11111 (full health) to 55555 (worst health). A lower score means a better outcome.
EuroQol 5-Dimension 5-Level (EQ-5D-5L) | three-month follow-up
  EuroQol 5-Dimension 5-Level (EQ-5D-5L), is the 5-digit code measuring functional ability. Each dimension in the EQ-5D-5L has five response levels: no problems (Level 1); slight; moderate; severe; and extreme problems (Level 5). There are 3,125 possible health states defined by combining one level from each dimension, ranging from 11111 (full health) to 55555 (worst health). A lower score means a better outcome.
36-item Short Form Health Survey (SF-36) | immediately before treatment 1
  36-item Short Form Health Survey (SF-36) measured functional ability. It has a two-step interpretation. First, precoded numeric values are recoded per the scoring key. Each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100. A high score means a better outcome. In step 2, items in the same scale are averaged together to create the 8 scale scores.
36-item Short Form Health Survey (SF-36) | one-month follow-up
  36-item Short Form Health Survey (SF-36) measured functional ability. It has a two-step interpretation. First, precoded numeric values are recoded per the scoring key. Each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100. A high score means a better outcome. In step 2, items in the same scale are averaged together to create the 8 scale scores.
36-item Short Form Health Survey (SF-36) | three-month follow-up
  36-item Short Form Health Survey (SF-36) measured functional ability. It has a two-step interpretation. First, precoded numeric values are recoded per the scoring key. Each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100. A high score means a better outcome. In step 2, items in the same scale are averaged together to create the 8 scale scores.
Barthel Index | immediately before treatment 1
  Barthel Index is a 10-item functional ability measure. An overall score is reached by adding the scores for each item and this ranges from 0 to 100. A higher score means a better outcome.
Barthel Index | one-month follow-up
  Barthel Index is a 10-item functional ability measure. An overall score is reached by adding the scores for each item and this ranges from 0 to 100. A higher score means a better outcome.
Barthel Index | three-month follow-up
  Barthel Index is a 10-item functional ability measure. An overall score is reached by adding the scores for each item and this ranges from 0 to 100. A higher score means a better outcome.
Change from Baseline Client Service Receipt Inventory | three-month follow-up
  Client Service Receipt Inventory will be used for assessing participants' socio-economic conditions without any scores calculated. No minimum and maximum values.
Work and Social Adjustment Scale | immediately before treatment 1
  Work and Social Adjustment Scale will be used to assess participants' socioeconomic conditions. Each item is rated on a 9-point scale from 0 (no impairment at all) to 8 (very severe impairment), so the total score is ranging from 0 to 40. Lower scores mean a better outcome.
Work and Social Adjustment Scale | one-month follow-up
  Work and Social Adjustment Scale will be used to assess participants' socioeconomic conditions. Each item is rated on a 9-point scale from 0 (no impairment at all) to 8 (very severe impairment), so the total score is ranging from 0 to 40. Lower scores mean a better outcome.
Work and Social Adjustment Scale | three-month follow-up
  Work and Social Adjustment Scale will be used to assess participants' socioeconomic conditions. Each item is rated on a 9-point scale from 0 (no impairment at all) to 8 (very severe impairment), so the total score is ranging from 0 to 40. Lower scores mean a better outcome.
Generalised Anxiety Disorder 7 (GAD-7) | immediately before treatment 1
  Generalised Anxiety Disorder 7 (GAD-7) will be used for evaluating participants' psychological conditions; scores from 0 to 21, higher scores mean a worse outcome.
Generalised Anxiety Disorder 7 (GAD-7) | one-month follow-up
  Generalised Anxiety Disorder 7 (GAD-7) will be used for evaluating participants' psychological conditions; scores from 0 to 21, higher scores mean a worse outcome.
Generalised Anxiety Disorder 7 (GAD-7) | three-month follow-up
  Generalised Anxiety Disorder 7 (GAD-7) will be used for evaluating participants' psychological conditions; scores from 0 to 21, higher scores mean a worse outcome.
Patient Health Questionnaire 9 (PHQ9) | immediately before treatment 1
  Patient Health Questionnaire 9 (PHQ9) will be used for evaluating participants' psychological conditions; scores from 0 to 27, higher scores mean a worse outcome.
Patient Health Questionnaire 9 (PHQ9) | one-month follow-up
  Patient Health Questionnaire 9 (PHQ9) will be used for evaluating participants' psychological conditions; scores from 0 to 27, higher scores mean a worse outcome.
Patient Health Questionnaire 9 (PHQ9) | three-month follow-up
  Patient Health Questionnaire 9 (PHQ9) will be used for evaluating participants' psychological conditions; scores from 0 to 27, higher scores mean a worse outcome.
Adapted Patient Health Questionnaire 15 (PHQ15) | immediately before treatment 1
  Adapted Patient Health Questionnaire 15 (PHQ15) will be used for evaluating participants' psychological conditions; scores from 0 to 30, higher scores mean a worse outcome.
Adapted Patient Health Questionnaire 15 (PHQ15) | one-month follow-up
  Adapted Patient Health Questionnaire 15 (PHQ15) will be used for evaluating participants' psychological conditions; scores from 0 to 30, higher scores mean a worse outcome.
Adapted Patient Health Questionnaire 15 (PHQ15) | three-month follow-up
  Adapted Patient Health Questionnaire 15 (PHQ15) will be used for evaluating participants' psychological conditions; scores from 0 to 30, higher scores mean a worse outcome.
Multiscale Dissociation Inventory (MDI) | immediately before treatment 1
  Multiscale Dissociation Inventory (MDI), a 30-item self-report test, evaluates participants' psychological conditions. It has a two-step interpretation. First, scoring each item using a scale ranging from 1 (never) to 5 (very often). In step 2, items in the same scale are summed together to create the 6 scale scores so the total score of each scale is from 5 to 25. A higher score means a worse outcome.
Multiscale Dissociation Inventory (MDI) | one-month follow-up
  Multiscale Dissociation Inventory (MDI), a 30-item self-report test, evaluates participants' psychological conditions. It has a two-step interpretation. First, scoring each item using a scale ranging from 1 (never) to 5 (very often). In step 2, items in the same scale are summed together to create the 6 scale scores so the total score of each scale is from 5 to 25. A higher score means a worse outcome.
Multiscale Dissociation Inventory (MDI) | three-month follow-up
  Multiscale Dissociation Inventory (MDI), a 30-item self-report test, evaluates participants' psychological conditions. It has a two-step interpretation. First, scoring each item using a scale ranging from 1 (never) to 5 (very often). In step 2, items in the same scale are summed together to create the 6 scale scores so the total score of each scale is from 5 to 25. A higher score means a worse outcome.
Emotion Regulation Questionnaire (ERQ) | immediately before treatment 1
  Emotion Regulation Questionnaire (ERQ), a 10-item scale designed to measure respondents' tendency to regulate their emotions in two ways: Cognitive Reappraisal (items 1, 3, 5, 7, 8, 10) and Expressive Suppression (items 2, 4, 6, 9). Respondents answer each item on a 7-point Likert-type scale ranging from 1 (strongly disagree) to 7 (strongly agree). The scoring takes the average of all the scores ranging from 1 to 7. Higher scores mean better outcomes.
Emotion Regulation Questionnaire (ERQ) | one-month follow-up
  Emotion Regulation Questionnaire (ERQ), a 10-item scale designed to measure respondents' tendency to regulate their emotions in two ways: Cognitive Reappraisal (items 1, 3, 5, 7, 8, 10) and Expressive Suppression (items 2, 4, 6, 9). Respondents answer each item on a 7-point Likert-type scale ranging from 1 (strongly disagree) to 7 (strongly agree). The scoring takes the average of all the scores ranging from 1 to 7. Higher scores mean better outcomes.
Emotion Regulation Questionnaire (ERQ) | three-month follow-up
  Emotion Regulation Questionnaire (ERQ), a 10-item scale designed to measure respondents' tendency to regulate their emotions in two ways: Cognitive Reappraisal (items 1, 3, 5, 7, 8, 10) and Expressive Suppression (items 2, 4, 6, 9). Respondents answer each item on a 7-point Likert-type scale ranging from 1 (strongly disagree) to 7 (strongly agree). The scoring takes the average of all the scores ranging from 1 to 7. Higher scores mean better outcomes.
Multidimensional Assessment of Interoceptive Awareness, version 2 (MAIA-2) | immediately before treatment 1
  Multidimensional Assessment of Interoceptive Awareness, version 2 (MAIA-2) is a self-report questionnaire with 37 items to measure interoception. It has a two-step interpretation. First, scoring each item on a six-point Likert scale from 0 (never) to 5 (always). In step 2, items in the same scale are averaged together to create the 8 scale scores. So the minimum score is 0 and the maximum score is 5. Higher scores mean a better outcome.
Multidimensional Assessment of Interoceptive Awareness, version 2 (MAIA-2) | one-month follow-up
  Multidimensional Assessment of Interoceptive Awareness, version 2 (MAIA-2) is a self-report questionnaire with 37 items to measure interoception. It has a two-step interpretation. First, scoring each item on a six-point Likert scale from 0 (never) to 5 (always). In step 2, items in the same scale are averaged together to create the 8 scale scores. So the minimum score is 0 and the maximum score is 5. Higher scores mean a better outcome.
Multidimensional Assessment of Interoceptive Awareness, version 2 (MAIA-2) | three-month follow-up
  Multidimensional Assessment of Interoceptive Awareness, version 2 (MAIA-2) is a self-report questionnaire with 37 items to measure interoception. It has a two-step interpretation. First, scoring each item on a six-point Likert scale from 0 (never) to 5 (always). In step 2, items in the same scale are averaged together to create the 8 scale scores. So the minimum score is 0 and the maximum score is 5. Higher scores mean a better outcome.
Sense of Agency Scale (SoAS) | immediately before treatment 1
  Sense of Agency scale (SoAS), a 13-item scale designed to measure respondents' sense of agency in two ways: Sense of Positive Agency (SoPA) and Sense of Negative Agency (SoNA). Respondents answer each item on a 7-point Likert-type scale ranging from 1 (totally disagree) to 7 (fully agree). The scoring takes the sum of all the scores so the minimum scores are 6 (SoPA) or 7 (SoNA) and the maximum scores are 42 (SoPA) or 49 (SoNA). Higher scores mean better outcomes.
Sense of Agency Scale (SoAS) | one-month follow-up
  Sense of Agency scale (SoAS), a 13-item scale designed to measure respondents' sense of agency in two ways: Sense of Positive Agency (SoPA) and Sense of Negative Agency (SoNA). Respondents answer each item on a 7-point Likert-type scale ranging from 1 (totally disagree) to 7 (fully agree). The scoring takes the sum of all the scores so the minimum scores are 6 (SoPA) or 7 (SoNA) and the maximum scores are 42 (SoPA) or 49 (SoNA). Higher scores mean better outcomes.
Sense of Agency Scale (SoAS) | three-month follow-up
  Sense of Agency scale (SoAS), a 13-item scale designed to measure respondents' sense of agency in two ways: Sense of Positive Agency (SoPA) and Sense of Negative Agency (SoNA). Respondents answer each item on a 7-point Likert-type scale ranging from 1 (totally disagree) to 7 (fully agree). The scoring takes the sum of all the scores so the minimum scores are 6 (SoPA) or 7 (SoNA) and the maximum scores are 42 (SoPA) or 49 (SoNA). Higher scores mean better outcomes.
Pittsburgh Sleep Quality Index (PSQI) | immediately before treatment 1
  Pittsburgh Sleep Quality Index (PSQI) will be used for assessing participants' sleep quality; scores from 0 to 21, higher scores mean a worse outcome.
Pittsburgh Sleep Quality Index (PSQI) | immediately before treatment 2
  Pittsburgh Sleep Quality Index (PSQI) will be used for assessing participants' sleep quality; scores from 0 to 21, higher scores mean a worse outcome.
Pittsburgh Sleep Quality Index (PSQI) | one-month follow-up
  Pittsburgh Sleep Quality Index (PSQI) will be used for assessing participants' sleep quality; scores from 0 to 21, higher scores mean a worse outcome.
Pittsburgh Sleep Quality Index (PSQI) | three-month follow-up
  Pittsburgh Sleep Quality Index (PSQI) will be used for assessing participants' sleep quality; scores from 0 to 21, higher scores mean a worse outcome.
Salivary cortisol | immediately before treatment 1
  Salivary cortisol will be measured to assess participants' stress
Salivary cortisol | immediately before treatment 2
  Salivary cortisol will be measured to assess participants' stress
Salivary cortisol | one-month follow-up
  Salivary cortisol will be measured to assess participants' stress
Actigraphy | baseline
  Actigraphy-derived level of activity will be analysed to measure participants' activities. It reports parameters of activities such as time, frequency.
Actigraphy | immediately after treatment 1
  Actigraphy-derived level of activity will be analysed to measure participants' activities. It reports parameters of activities such as time, frequency.
Actigraphy | immediately before treatment 2
  Actigraphy-derived level of activity will be analysed to measure participants' activities. It reports parameters of activities such as time, frequency.
Adverse events (AE) | immediately before treatment 1
  Adverse events details will be recorded
Adverse events (AE) | immediately after treatment 1
  Adverse events details will be recorded
Adverse events (AE) | immediately before treatment 2
  Adverse events details will be recorded
Adverse events (AE) | immediately after treatment 2
  Adverse events details will be recorded
Adverse events (AE) | one-month follow-up
  Adverse events details will be recorded
Adverse events (AE) | three-month follow-up
  Adverse events details will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Nicholson, MBBS, PhD, Principal Investigator — King's College London
Locations (1):
- Institute of Psychiatry, Psychology & Neuroscience, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Personally identifiable or sensitive individual participant data will not be shared to protect the participants' confidentiality.